CLINICAL TRIAL: NCT02523729
Title: Effects of Anke Malz on Women During Lactation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: Lorillard Tobacco Company (Industry)
Responsible Party: Principal Investigator, Hui-Ting Yang, associate professor, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CMUH102-REC3-053
Record Dates: First submitted 2015-03-03; First posted 2015-08-14 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Non-alcoholic Malt Product in Lactation
Keywords: lactation; human milk; maltz; antioxidant
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- control (No Intervention): subjects drunk no Anke Malz product.
- intervention one (Experimental): subjects drunk one can Anke Malz product.
  Interventions: Dietary Supplement: Anke Malz
- intervention two (Experimental): subjects drunk two cans Anke Malz product.
  Interventions: Dietary Supplement: Anke Malz

INTERVENTIONS:
Dietary Supplement: Anke Malz — non-alcoholic malt drink
  Arms: intervention one; intervention two

SUMMARY:
Human milk is the most optimal food to provide all infants' needs before eating solid food. However, underproduction of milk is a common and concerned problem for breastfeeding women. In this case, proper milk-making foods reveal their importance on lactation. In many European countries, ancient wisdom clams that non-alcoholic malt beverage could facilitate the secretion of breast milk. This study estimates the effects of non-alcoholic malt product during first three months of lactation.

ELIGIBILITY:
Inclusion Criteria:

* Single fetal pregnancy
* Full time birth

Exclusion Criteria:

* Any complication during pregnancy
* Smokers
* Alcohol or drug abuse

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
The concentration of prolactin on lactational women | three months

SECONDARY OUTCOMES:
Mean breast-feeding time | three months

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ting Yang, Doctor, Study Chair — Department of Nutrition, China Medical University, Taiwan

REFERENCES:
- [Background] Grossman ER. Beer, breast-feeding, and the wisdom of old wives. JAMA. 1988 Feb 19;259(7):1016. No abstract available. PMID 3339797
- [Result] Foo LL, Quek SJ, Ng SA, Lim MT, Deurenberg-Yap M. Breastfeeding prevalence and practices among Singaporean Chinese, Malay and Indian mothers. Health Promot Int. 2005 Sep;20(3):229-37. doi: 10.1093/heapro/dai002. Epub 2005 Apr 6. PMID 15814526
- [Result] Carlson HE, Wasser HL, Reidelberger RD. Beer-induced prolactin secretion: a clinical and laboratory study of the role of salsolinol. J Clin Endocrinol Metab. 1985 Apr;60(4):673-7. doi: 10.1210/jcem-60-4-673. PMID 3972968
- [Result] Ballard O, Morrow AL. Human milk composition: nutrients and bioactive factors. Pediatr Clin North Am. 2013 Feb;60(1):49-74. doi: 10.1016/j.pcl.2012.10.002. PMID 23178060
- [Result] Adiong JP, Kim E, Koren G, Bozzo P. Consuming non-alcoholic beer and other beverages during pregnancy and breastfeeding. Can Fam Physician. 2014 Aug;60(8):724-5. PMID 25122816